CLINICAL TRIAL: NCT05719311
Title: SPAN: A Phase 2, Open Label, Multicenter, Pilot Study to Assess Safety and Efficacy of an Enteric Microgranule Formulation of Adrulipase in Patients With Exocrine Pancreatic Insufficiency (EPI) Due to Cystic Fibrosis (CF)
Brief Title: Study to Assess an Enteric Microgranule Formulation of Adrulipase in Patients With Cystic Fibrosis
Acronym: SPAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Entero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FWB-CF-2.03
Record Dates: First submitted 2023-01-31; First posted 2023-02-08 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-07

CONDITIONS: Exocrine Pancreatic Insufficiency; Cystic Fibrosis
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Adrulipase (Experimental): Upon study enrolment, the patient will be switched from their commercial PERT to receive adrulipase. Patients will initially receive a low dose of adrulipase. Upon the appearance of EPI symptoms, lasting at least three days, and upon discussion with the investigator, the patient will be switched to the medium dose of adrulipase. If signs and symptoms of EPI persist for three or more days, the patient will be switched to the high dose of adrulipase.
  Interventions: Drug: adrulipase

INTERVENTIONS:
Drug: adrulipase — Enteric microgranule formulation of adrulipase.
  Other Names: MS1819

SUMMARY:
Some cystic fibrosis patients are unable to digest food and absorb nutrition appropriately as they have a condition known as exocrine pancreatic insufficiency (EPI). Currently, these patients take pancreatic enzymes that are obtained from pig pancreas to aid the digestion of food. The goals of this clinical study are to evaluate the safety and efficacy of a novel formulation of a non-porcine lipase, called adrulipase, in patients with EPI due to cystic fibrosis.

The main question[s] the study aims to answer are:

1. Is the novel formulation of adrulipase safe to use at the doses being evaluated in the clinical study.
2. Is adrulipase as effective, or more effective, compared to the pig enzymes the patients currently use.

Researchers will compare the results obtained with adrulipase to how the patients typically respond to their pig enzymes to see if adrulipase helps patients digest fats adequately and if their stomach feels good (signs and symptoms of malabsorption).

DETAILED DESCRIPTION:
This is an Phase 2, open label, single arm pilot study assessing the safety and efficacy of adrulipase in an enteric microgranule formulation. Patients with a confirmed diagnosis of cystic fibrosis who are 18 years of age or greater will be screened for eligibility if they have been clinically controlled on a stable dose of commercial pancreatic enzyme replacement therapy (PERT) for at least one month. Patients on cystic fibrosis transmembrane conductance regulator (CFTR) modulator therapies must have been on a stable dose for at least 3 months prior to study entry, and no dose changes will be made during the study. Patients receiving gastric acid suppressants must have been on a stable dose for at least one month prior to study entry and no dose changes will be made during the study.

Upon obtaining an informed consent, potentially eligible patients will receive dietary counselling during the week prior to the scheduled date of confinement for collecting stool samples for calculation of baseline coefficient of fat absorption (CFA). This counselling will emphasize the importance of dietary stability during the study. Patients found to have a CFA of 80% or greater while receiving their commercial PERT and meeting the other eligibility criteria will be enrolled into the study.

Upon study enrolment, the patient will be switched from their commercial PERT to receive adrulipase. The patient will remain on study for approximately three weeks, after which a repeat CFA will be obtained. A dose titration scheme will be used for determining whether a low, medium, or high dose of adrulipase may succeed in controlling signs and symptoms of exocrine pancreatic insufficiency (EPI) and provide a CFA of 80% or greater. Patients will initially receive a low dose of adrulipase. Upon the appearance of EPI symptoms, lasting at least three days, and upon discussion with the investigator, the patient will be switched to the medium dose of adrulipase. If signs and symptoms of EPI persist for three or more days, the patient will be switched to the high dose of adrulipase. After patients reach 3 weeks of study and complete their end of study CFA, they will be returned to their pre-study commercial PERT. An end of study safety visit will be scheduled for one week after finishing adrulipase therapy.

Safety assessments will be made by collecting adverse events, safety lab assessments, and immunologic assays to assess drug induced immune responses.

ELIGIBILITY:
Inclusion Criteria:

1. A confirmed diagnosis of cystic fibrosis, based on 2 clinical features consistent with CF, plus either a new/historic sweat chloride >60 mmol/L by quantitative pilocarpine iontophoresis (measured while not on a CFTR modulator) or genotype.
2. On stable dose of porcine PERT ≥1 month (30 days) prior to screening; stable dose is defined as dose of medication not changed during this time period, and the medication must be commercially available and be administered in the recommended dose range.
3. CFA = or > 80% at screening while on stable PERT
4. A fair or better nutritional status as defined by:

   * BMI ≥16.0 kg/m2 for female patients ≥18 years of age, or
   * BMI ≥16.5 kg/m2 for male patients ≥18 years of age
5. Fecal elastase <100 µg/g of stool at screening
6. Standard-of-Care medications including CFTR modulators are allowed

Exclusion Criteria:

1. History or diagnosis of fibrosing colonopathy
2. Any chronic diarrheal illness unrelated to pancreatic insufficiency
3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level

   * 5 ×upper limit of normal (ULN), or total bilirubin level ≥1.5 ×ULN at Screening
4. Feeding via an enteral tube during 6 months before screening
5. Forced expiratory volume ≤30% at the Screening visit
6. Changes in gastric acid suppressant therapy during the one month prior to screening for patients already on suppressant therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Central Florida Pulmonary Group, Orlando, Florida
  - The Cystic Fibrosis Institute, Northfield, Illinois
  - Childrens Lung Specialists, Las Vegas, Nevada

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adrulipase
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Adrulipase
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Safety of Adrulipase
Description: Number of subjects reporting 1 or more adverse events.
Time Frame: End of 3-week treatment period.
Measure: Count of Participants; unit: Participants
Groups:
- Adrulipase: Adrulipase
Arm/Group | Adrulipase
Number analyzed (Participants) | 13
Participants | 2

2. Primary Outcome: Efficacy of Adrulipase: Coefficient of Fat Absorption (CFA)
Description: The primary efficacy endpoint is the CFA that will be assessed at the end of the 3-week treatment period. CFAs for adrulipase will be compared to the CFAs of PERT obtained at baseline/eligibility using descriptive methods.
Time Frame: End of 3-week treatment period.
Population: Number of participants that achieved a CFA >= 80%
Measure: Count of Participants; unit: Participants
Arm/Group | Adrulipase
Number analyzed (Participants) | 13
Participants | 2

3. Secondary Outcome: Stool Weight
Description: Stool weights obtained during the supervised confinement visit at the end of the 3-week treatment period will be measured. Stool weights obtained during confinement on adrulipase will be compared to the stool weights during confinement on PERT obtained at baseline/eligibility using descriptive methods.
Time Frame: Change between two time points: initial PERT confinement and end of 3-week treatment period.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Adrulipase
Number analyzed (Participants) | 13
grams | 647.1 (496.41)

4. Secondary Outcome: Coefficient of Nitrogen Absorption (CNA)
Description: CNA that will be assessed at the end of the 3-week treatment period. CNAs for adrulipase will be compared to the CNAs of PERT obtained at baseline/eligibility using descriptive methods.
Time Frame: Change between two time points: initial PERT confinement and end of 3-week treatment period
Measure: Mean (Standard Deviation); unit: Percentage of nitrogen absorbed
Arm/Group | Adrulipase
Number analyzed (Participants) | 13
Percentage of nitrogen absorbed | -27.8 (14.47)

ADVERSE EVENTS:
Time Frame: 3-weeks
Groups:
- Low Dose: Adrulipase (1.95 g/day)
- Mid Dose: Adrulipase (2.4 g/day)
- High Dose: Adrulipase (3.3 g/day)
Arm/Group | Low Dose | Mid Dose | High Dose
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/5 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/1 | 2/5 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose (N=1) | Mid Dose (N=5) | High Dose (N=7)
Unclear etiology (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT05719311/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/11/NCT05719311/SAP_001.pdf